CLINICAL TRIAL: NCT00271414
Title: A 15-day Trial to Document the Safety, Clinical Utility and Pharmacokinetics of Duragesic (TTS Fentanyl) in the Treatment of Pediatric Subjects With Continuous Pain Requiring Opioid Therapy
Brief Title: A 15-day Study to Assess the Safety and Clinical Utility of Duragesic (Fentanyl Transdermal Patch) in the Treatment of Children With Continuous Pain Requiring Narcotic Pain Relief Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005962
Record Dates: First submitted 2005-12-30; First posted 2006-01-02 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Pain
Keywords: chronic pain; opioid; fentanyl; transdermal; Duragesic; morphine
MeSH Terms: conditions — Chronic Pain | interventions — Fentanyl

INTERVENTIONS:
Drug: Duragesic® (fentanyl) Transdermal Therapeutic System (TTS)

SUMMARY:
The objective of this study is to assess the safety and clinical utility of DuragesicÂ® 12.5 micrograms/hour (a transdermal patch delivering the narcotic pain-reliever fentanyl) in the treatment of children ages 2 to 12 with continuous pain requiring narcotic pain relief therapy. Pharmacokinetics (fentanyl levels in the bloodstream during treatment) will also be assessed.

DETAILED DESCRIPTION:
A new dosage strength of Duragesic® TTS patch was developed to deliver 12.5 micrograms of fentanyl per hour, which is considered to be equi-analgesic to a daily dose of 45 mg of morphine administered orally, and considered a safe starting dose in children aged 2 to 12 years. This is a single-arm, non-randomized, open-label, 15-day multicenter trial to determine the safety, clinical utility, and pharmacokinetics of Duragesic® in pediatric subjects who require treatment with a potent opioid for the management of continuous pain, allowing individual titration. After the 15-day primary treatment period, subjects may, at the investigator's discretion, continue long-term treatment with Duragesic® for a period of up to 1 year.

All subjects start treatment with a 12.5 micrograms/hour patch. Immediate-release morphine is available to treat breakthrough pain. The patches are replaced every 72 hours. The objective is to have subjects pain-free as much as possible, using the least possible rescue medication. Duragesic® dose increases are considered based on rescue medication consumption and pain assessment. Where a subject is maintained pain-free with a daily consumption of 45 mg of rescue morphine or more, a dose increase of Duragesic® with 12.5 micrograms/hour is permitted. No increase in Duragesic® dose is to be performed within the 72-hour dosing interval. The primary outcome of this study is an assessment of safety, including the incidence and severity of adverse events, and physical examination results and vital signs. Clinical utility is assessed by the parent's treatment assessment of pain relief, tolerability and convenience (pre-treatment and after each patch change); the investigator's and the parent's global assessments on Day 16 of pain control, adverse events, and convenience; daily measures of pain levels; use of rescue medication; and the child's play performance. Pharmacokinetics will also be assessed. Duragesic® will be applied to the upper torso, and replaced every 72 hours. The initial dose is one patch with a fentanyl delivery rate of approximately 12.5 micrograms/hour. Dose increases in steps of 12.5 micrograms/hour are considered if pain is inadequately controlled. The treatment phase is 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric (age 2-12) patients suffering from continuous pain of a well-documented cause
* currently requiring treatment of pain with a strong opioid and expected to continue to require treatment with a strong opioid for the next 7 days
* prior therapy for pain included a minor analgesic, weak opioid, or strong opioid equivalent to the pain relief of 45 mg morphine or less a day

Exclusion Criteria:

* Patients with a history of allergy or hypersensitivity to fentanyl or morphine
* have active skin disease that precludes application of Duragesic® or which may affect the absorption of fentanyl
* have a life expectancy was less than 1 month
* have a clinical condition that in the investigator's judgment prevents participation in the study (e.g., clinically relevant liver dysfunction), plan to undergo a surgical procedure within 3 days of study entry, or are currently using protease inhibitors (HIV/AIDS treatment)
* have participated in any other drug trial relating to pain control within one month of study entry or currently participating in any other study or research project which would interfere with this trial

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 1999-03; Study Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events; Physical examination results and vital signs; Pharmacokinetics

SECONDARY OUTCOMES:
Parent's assessment of pain relief, tolerability and convenience (pre-treatment and after patch changes); Investigator's/parent's global assessments on Day 16 of pain control, adverse events, and convenience; Daily pain levels; Rescue medication usage

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- See also: A 15-day study to assess the safety and clinical utility of Duragesic� (fentanyl transdermal patch) in the treatment of children with continuous pain requiring narcotic pain relief therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=390&filename=CR005962_CSR.pdf